CLINICAL TRIAL: NCT05855135
Title: Assessment of the Safety and Efficacy of a Combined Cardiac Contractility Modulation and Implantable Cardioverter Defibrillator Device for Subjects With Heart Failure and Reduced Ejection Fraction
Brief Title: Assessment of Combined CCM and ICD Device in HFrEF
Acronym: INTEGRA-D
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Impulse Dynamics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG_PRO_345
Record Dates: First submitted 2023-05-03; First posted 2023-05-11 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure; Heart Failure With Reduced Ejection Fraction; Implantable Defibrillator User; CCM Therapy; Non-ischemic Cardiomyopathy; Ischemic Cardiomyopathy; Sudden Cardiac Arrest; Arrhythmias, Cardiac; Ventricular Tachycardia; Ventricular Fibrillation
Keywords: Heart Failure; HFrEF; Stage C Heart Failure; Stage D Heart Failure; Defibrillation Efficacy Testing; Induced Ventricular Fibrillation; Ventricular fibrillation; Ventricular tachycardia; Implantable cardioverter defibrillator; Sudden cardiac arrest
MeSH Terms: conditions — Heart Failure; Death, Sudden, Cardiac; Arrhythmias, Cardiac; Tachycardia, Ventricular; Ventricular Fibrillation

STUDY DESIGN:
Intervention Model Description: Single arm, prospective, multicenter study of 300 subjects that will establish that the device can appropriately sense and convert episodes of induced VF "on the table" in the implant procedure room, spontaneous episodes of VT/VF that occur during the study follow-up period, and ensure that the inappropriate shock rate is not unacceptably high.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- CCM-D Implant (Experimental): The subject is implanted with the CCM-D device.
  Interventions: Device: OPTIMIZER® Integra CCM-D System (Treatment Arm)

INTERVENTIONS:
Device: OPTIMIZER® Integra CCM-D System (Treatment Arm) — The CCM-D System is an implantable cardiac device system that combines cardiac contractility modulation and implantable cardioverter defibrillator (ICD) modules into one device. CCM-D is also known as a "Cardiac Contractility Modulation - Defibrillator". All 300 subjects will be implanted with the CCM-D System and followed for a period of at least two years.

SUMMARY:
The goal of this clinical trial is to demonstrate that the OPTIMIZER® Integra CCM-D System (the "CCM-D System") can safely and effective convert induced ventricular fibrillation (VF) and spontaneous ventricular tachycardia and/or ventricular fibrillation (VT/VF) episodes in subjects with Stage C or D heart failure who remain symptomatic despite being on guideline-directed medical therapy (GDMT), are not indicated for cardiac resynchronization therapy (CRT), and have heart failure with reduced left ventricular ejection fraction (LVEF ≤40%).

Eligible subjects will be implanted with the CCM-D System. A subset of subjects will be induced into ventricular fibrillation "on the table" in the implant procedure room. During the follow-up period, inappropriate shock rate and device-related complications will be evaluated. The follow-up period is expected to last at least two years.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all the following:

1. Patient is aged 18 years or older;
2. Patient meets the Stage C or D criteria of the Universal Definition of Heart Failure ;
3. Patient has HFrEF (LVEF ≤40%);
4. Patient is on GDMT for heart failure;
5. Patient has a Class I or Class II indication for an ICD
6. Patient has a reasonable expectation of meaningful survival of > 1 year;
7. Patient has either non-ischemic cardiomyopathy or ischemic cardiomyopathy and is at least 40 days post-MI, if an MI occurred;
8. Patient is willing to give informed consent, available for scheduled study follow-up visits, and able to complete all testing described in the study protocol at the investigational site location.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Patients should not have severe AI or AS, and should not have MS; additionally, patients undergoing DE testing should not have severe MR;
2. Patients who have undergone mitral valve repair or clip within 90 days prior to study consent;
3. Cardiac surgery within 90 days or a PCI procedure within 30 days prior to study consent;
4. Prior heart transplant or ventricular assist device;
5. Implanted mechanical tricuspid valve;
6. PR interval greater than 375ms or advanced AV block;
7. In situ S-ICD, pacemaker, or CRT device;
8. Indicated for CRT;
9. End stage renal disease, currently on dialysis, or with other major medical disorder (e.g. liver failure, terminal cancer);
10. Indicated for permanent bradyarrhythmia pacing;
11. Unstable angina pectoris within 30 days prior to study consent;
12. Pregnant or planning to become pregnant during the study;
13. Participating in another cardiac investigational device or drug study at the same time (or within 30 days prior to study consent); Note: Registries and other observational studies are acceptable.
14. Other criteria that preclude Optimizer INTEGRA CCM-D implantation and/or CCM therapy, as determined by Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-17 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Device Effectiveness in Converting Induced Ventricular Fibrillation (Primary Efficacy Objective) | Implant
  Evaluate the device effectiveness in converting induced VF at the time of implantation.
Device-related Complications (Primary Safety Objective) | Implant to 6 months
  Evaluate device-related complications through 6-months (excluding lead-related complications).

SECONDARY OUTCOMES:
Inappropriate Shock Rate out to 6-months (Secondary Safety Objective) | Implant to 6 months
  Evaluate the incidence of inappropriate ICD shocks through the time when the last subject enrolled completes the 6-month visit.

OTHER OUTCOMES:
Inappropriate Shock Rate out to 2-years | Implant to 2 years
  Evaluate the device effectiveness in converting spontaneous VT/VF through the time when the last subject enrolled completes the 6-month visit. Each subject will be followed for 2-years after implant to capture additional spontaneous episodes that may occur.
Charging non-compliance | Implant to 2 years
  Evaluate subject charging non-compliance defined as >14 days between interval charging sessions, overall and frequency of non-compliance in the same subject.
Longitudinal levels of activity | Implant to 2 years
  Track longitudinal levels of activity weekly via OPTIhome (when available) and identification of trends.
Battery degradation and longevity | Implant to 2 years
  Assess battery degradation and longevity either remotely or during an in-person follow-up at 2 years (+/- 60 days) by recording QHR battery voltage as measured by the Integra CCM-D IPG. The measurement under nominal conditions is expected to be 2.85V or higher, consistent with a 20-year device longevity.
Compare worsening heart failure events pre- and post-implant | 12 months prior to implant and 12 months post-implant
  Track unscheduled cardiovascular-related healthcare encounters from 12 months prior to implant, if available, to 12 months post-implant
All-cause mortality | 1 and 2 years post-implant
  Assess all-cause mortality using Seattle Heart Failure Model (SHFM) and comorbidity burden as a predictive comparator at 1 year and 2 years post-implant
Kansas City Cardiomyopathy Questionnaire (KCCQ) | Baseline to 6-months
  Compare change in subject's perception of their heart failure symptoms, as measured by KCCQ, from baseline to 6 months.
EQ-5D-5L | Baseline to 6-months
  Compare change in subject's perception of their health status, as measured by the EQ-5D-5L, from baseline to 6 months.
Six Minute Walk Distance (6MWD) | Baseline to 6 months
  Compare change in functional capacity, as measured by 6MWD, from baseline to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Varma, MD, PhD, Principal Investigator — The Cleveland Clinic; Nir Uriel, MD, Principal Investigator — Columbia University
Locations (59):
- United States (59):
  - Phoenix Heart, Glendale, Arizona
  - CardioVascular Associates of Mesa, Mesa, Arizona
  - Southwest Cardiovascular Associates, Mesa, Arizona
  - Arizona Heart Rhythm, Phoenix, Arizona
  - CVC Cardiovascular Consultants, Phoenix, Arizona
  - Phoenix Heart, Phoenix, Arizona
  - Honor Health, Scottsdale, Arizona
  - University of Southern California, Los Angeles, California
  - Cedars Sinai Medical Center, Los Angeles, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - Hartford HealthCare, Hartford, Connecticut
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Baptist Health South Florida, Miami, Florida
  - Mount Sinai Medical Center Miami Beach, Miami Beach, Florida
  - Advent Health Orlando, Orlando, Florida
  - Cleveland Clinic Weston, Weston, Florida
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Baptist Health Lexington, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Saint Luke's Hospital, Kansas City, Missouri
  - St. Louis VA, St Louis, Missouri
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Virtua, Cherry Hill, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - The Heart House - Cardiovascular Associates of the Delaware Valley, Haddon Heights, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - NYU Langone, New York, New York
  - Mount Sinai New York, New York, New York
  - Columbia University Medical Center / NewYork-Presbyterian, New York, New York
  - Weill Cornell Medicine, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Sanger Heart and Vascular Institute, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - St. Francis Tulsa, Tulsa, Oklahoma
  - Portland VA Medical Center, Portland, Oregon
  - St. Luke's Bethlehem, Bethlehem, Pennsylvania
  - Bryn Mawr Medical Specialists Association, Bryn Mawr, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Penn Presbyterian, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Texas Cardiac Arrhythmia Research Foundation, Austin, Texas
  - Medical City Dallas, Dallas, Texas
  - UT Southwestern, Dallas, Texas
  - Medical City Fort Worth, Fort Worth, Texas
  - Houston Methodist, Houston, Texas
  - Houston VA Hospital, Houston, Texas
  - Christus Trinity Clinic, Tyler, Texas
  - Centra Health, Lynchburg, Virginia
  - Chippenham Hospital, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Seattle VA, Seattle, Washington
  - Swedish, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No